CLINICAL TRIAL: NCT03379324
Title: A Prospective, Randomized Study Comparing Outcomes Following Arthroscopic Double-row Rotator Cuff Repair With and Without the Addition of a Cryopreserved, Liquid, Injectable Amnion Allograft
Brief Title: Efficacy of an Amniotic Fluid Derived Allograft, (FlōGraft®) in Rotator Cuff Repairs: A Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Applied Biologics, LLC (Industry)
Collaborators: Fondren Orthopedic Group L.L.P. (Other); Texas Orthopedic Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOH169
Record Dates: First submitted 2017-11-20; First posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Rotator Cuff Tear; Fatty Atrophy
Keywords: Rotator Cuff; Human Amniotic Fluid; Amniotic Fluid Allograft; FlōGraft®; Amniotic Fluid Biologic; Fatty Atrophy; Fat Degeneration
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: This will be a stratified, randomized, radiograph and patient blinded, prospective trial enrolling 260 subjects undergoing rotator cuff repair
Who Masked: Participant, Outcomes Assessor
Masking Description: Eligible patients will be randomized to FlōGraft®-augmented repair versus repair alone. Surgeons cannot be blinded to treatment; however, follow-up MRIs will be assessed by blinded radiologists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superiority of augmented repairs (Active Comparator): Assess pain, function, and structural integrity of the rotator cuff at 3 months, 6 months, 1 year, and 2 years post-operation
  Interventions: Biological: Superiority of augmented repairs; Biological: Fat degeneration of supraspinatus muscle
- Fat degeneration of supraspinatus muscle (Active Comparator): MRI assessment the quantity and disposition of fat within the supraspinatus muscle body compared to pre-operation MRI, at 1 year and 2 years post-operation
  Interventions: Biological: Superiority of augmented repairs; Biological: Fat degeneration of supraspinatus muscle

INTERVENTIONS:
Biological: Superiority of augmented repairs — 4cc of FlōGraft® injected into repair subject tissue divided evenly between repair site and muscle body
  Other Names: FlōGraft®; Human amniotic fluid-derived allograft
Biological: Fat degeneration of supraspinatus muscle — 4cc of FlōGraft® injected into repair subject tissue divided evenly between repair site and muscle body
  Other Names: FlōGraft®; Human amniotic fluid-derived allograft

SUMMARY:
Rotator Cuff (RC) repair will be augmented with the injection of a human amniotic fluid derived allograft at the repair interface junction. A secondary injection will be administered at the time of repair in the supraspinatus muscle body medial to the musculotendonous junction.

DETAILED DESCRIPTION:
Patients will be given a written explanation of the study and screened for inclusion and exclusion criteria. Included patients will have a repairable, full thickness rotator cuff tear limited to the supraspinatus and infraspinatus, confirmed by MRI. Patients with concomitant biceps tenotomy, tenodesis, arthroscopic subacromial decompression, and distal clavicle excision will be included. Patients with prior operations on the shoulder, partial thickness tears, subscapularis tears or labral tears requiring repair, irreparable supraspinatus tears, staged bilateral rotator cuff repairs, or concomitant suprascapular nerve decompression will be excluded. We will also exclude patients with co-morbid conditions requiring the use of corticosteroids. Patients who cannot have an MRI for medical reasons will also be excluded.

All participants will volunteer to enroll in the study by signing informed consent (Attachment B). All potential subjects will be over 18 years of age and capable of providing their own informed consent. Patients will be recruited from the patient populations of Dr. Edwards, Dr. Elkousy, Dr. Morris, Dr. Gombera and Dr Brown. The informed consent process will be conducted by the investigators, their staff, or their research associates (e.g., orthopedic surgery fellows), who will explain the purpose and methods of the study, the risks and benefits, and requirements of participation. Randomization to groups will occur following informed consent; patients will not know to which group they are assigned.

1. Arthroscopic transosseous equivalent rotator cuff (TOE) repair will be performed; this is our standard procedure, using suture anchors in the medial and lateral rows for a TOE technique. The medial row will be 4.5 mm Polyether ether ketone (PEEK) anchors and the lateral row will be a 5.5 mm PEEK knotless anchor. Medial row anchor sutures will be tied.
2. FlōGraft® details: 4cc of FlōGraft® will be used in each treated patient, provided in a single peel pouch containing two 2cc vials. In FlōGraft® treated patients, FlōGraft® will be applied, following repair as detailed below.
3. FlōGraft® Preparation Protocol 3.1 Store FlōGraft® at -65◦C or colder until immediately prior to use. 3.2 Remove box from cold storage, open exterior box and remove interior package containing vials.

   3.3 Neither the interior dust cover nor the outside of the vial are sterile. Do not place either the interior package or the vial in sterile field.

   3.4 Remove vials from packaging, place on non-sterile, secure, flat surface, or hold vial firmly in one hand allowing contents to thaw (3-7 minutes.) Hold vial upright to aspirate contents. Note: Allograft should be implanted immediately post-thaw, but not later than eight (8) minutes post-thaw.

   3.5 Pierce the vial cap and draw thawed solution into syringe. Do not pressurize vial with air prior to extracting thawed FlōGraft® solution.

   3.6 If needed, change needle size based on surgeon preference (18g to 23g.)
4. FlōGraft® Implantation 4.1 After the rotator cuff repair is completed, shut off water-flow to joint. Excess water in joint is drained through the skin incisions, creating a "dry" sub-acromial space.

   4.2 Insert needle through skin incision or percutaneously. Under direct visualization, inject FlōGraft® directly into rotator cuff tissue at repair site in approximately 0.50 cc aliquots. Cover entire repair site.

   4.3 Implant allograft into the cuff muscle more medially to the repair in 0.25-0.5 cc aliquots, as appropriate.
5. Postoperative management: 4 weeks immobilization in abduction sling; passive range of motion will be initiated at the discretion of the surgeon based on tear size. Active range of motion will begin at 8 weeks to 16 weeks.
6. Diagnostic MRI will be performed at one and two years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Included patients will have a repairable, full thickness rotator cuff tear limited to the supraspinatus and infraspinatus, confirmed by MRI. Patients with concomitant biceps tenotomy, tenodesis, arthroscopic subacromial decompression, and distal clavicle excision will be included.

Exclusion Criteria:

* Patients with prior operations on the shoulder, partial thickness tears, subscapularis tears or labral tears requiring repair, irreparable supraspinatus tears, staged bilateral rotator cuff repairs, or concomitant suprascapular nerve decompression will be excluded. We will also exclude patients with co-morbid conditions requiring the use of corticosteroids. Patients who cannot have an MRI for medical reasons will also be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2017-03-24 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Structural healing integrity | 1 year post-operation
  Improved structural healing is the best indication of long-term surgery success. The Sugaya grading system is a method to account for structural integrity of the rotator cuff following surgery with five possible classifications. Sugaya scale: type I indicating sufficient thickness with homogeneously low intensity; type II, sufficient thickness with partial high intensity; type III, insufficient thickness without discontinuity; type IV, the presence of a minor discontinuity; and type V, the presence of a major discontinuity. Types I-III indicate different levels of healing. The classification of each shoulder must be assessed using MRIs (grade determined by a blinded musculoskeletal radiologist).

SECONDARY OUTCOMES:
Fatty degeneration | 1 year post-operation
  Musculoskeletal radiologists will also evaluate fatty degeneration of the rotator cuff at 1 year post-operatively from the MRI using the Global Fatty Degeneration Index (GFDI).
Structural healing integrity (2) | 2 years post-operation
  Improved structural healing is the best indication of long-term surgery success. The Sugaya grading system is a method to account for structural integrity of the rotator cuff following surgery with five possible classifications. Sugaya scale: type I indicating sufficient thickness with homogeneously low intensity; type II, sufficient thickness with partial high intensity; type III, insufficient thickness without discontinuity; type IV, the presence of a minor discontinuity; and type V, the presence of a major discontinuity. Types I-III indicate different levels of healing. The classification of each shoulder must be assessed using MRIs (grade determined by a blinded musculoskeletal radiologist).
Fatty degeneration (2) | 2 years post-operation
  Musculoskeletal radiologists will also evaluate fatty degeneration of the rotator cuff at 2 years post-operatively from the MRI using the Global Fatty Degeneration Index (GFDI).
Functional outcome | Baseline
  Functional outcomes will be assessed using the American Shoulder and Elbow Surgeons Score.
Functional outcome (2) | 3 months post-operation
  Functional outcomes will be assessed using the American Shoulder and Elbow Surgeons Score.
Functional outcome (3) | 6 months post-operation
  Functional outcomes will be assessed using the American Shoulder and Elbow Surgeons Score.
Clinically Assessed Re-tear | 3 months post-operation
  Any incidence of clinically assessed re-tear will be documented by the treating surgeon during routine postoperative follow-up clinic visits and examinations.
Clinically Assessed Re-tear (2) | 6 months post-operation
  Any incidence of clinically assessed re-tear will be documented by the treating surgeon during routine postoperative follow-up clinic visits and examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Stocks, MD, Study Chair — Texas Orthopedic Hospital
Locations (1):
- Texas Orthopedic Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No